CLINICAL TRIAL: NCT06041178
Title: Efficiency of Flurbiprofen 2.5% in Comparison to 98% Aloe Vera Gel as an Adjunctive Therapy to Scaling and Root Planning in the Initial Treatment of Stage III Chronic Periodontitis in Smoking Patients
Brief Title: Flurbiprofen Versus Aloe Vera Gel in the Treatment of Chronic Periodontitis in Smoking Patients.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Beirut Arab University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 2022-H-0100-D-R-0487
Record Dates: First submitted 2023-09-11; First posted 2023-09-18 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-08

CONDITIONS: Periodontitis Chronic Generalized Severe
MeSH Terms: interventions — Flurbiprofen

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- scaling and root planing + 2.5% flurbiprofen on one site and placebo on contralateral site (Experimental): Following scaling and root planing, the prepared 2.5% flurbiprofen was injected subgingivally in the selected deep pocket and the same was done with a placebo on the contralateral site
  Interventions: Drug: 2.5% flurbiprofen; Other: Placebo
- scaling and root planing + 98% aloe vera on one site and placebo on contralateral site (Experimental): Following scaling and root planing, the prepared aloe vera was injected subgingivally in the selected deep pocket and the same was done with a placebo on the contralateral site
  Interventions: Drug: 98% aloe vera; Other: Placebo
- scaling and root planing + 2.5% flurbiprofen on one site and 98% aloe vera on contralateral site (Experimental): Following scaling and root planing, the prepared 2.5% flurbiprofen was injected subgingivally in the selected deep pocket while the same was done with 98% aloe vera on the contralateral site
  Interventions: Drug: 2.5% flurbiprofen; Drug: 98% aloe vera

INTERVENTIONS:
Drug: 2.5% flurbiprofen — Gel was made of 20% poloxamer and 10% ethanol as an Optimum formulation with sustained release up to 48 hours and a reasonable sol gel transition phase (adjunctive to SRP)
  Arms: scaling and root planing + 2.5% flurbiprofen on one site and 98% aloe vera on contralateral site; scaling and root planing + 2.5% flurbiprofen on one site and placebo on contralateral site
Drug: 98% aloe vera — the Aloe vera gel employed possessed a concentration of 98% and was obtained from the reputable brand Avivir (Denmark). The remaining 2% comprised normal saline. The process of obtaining the 98% Aloe vera gel involved meticulous washing of mature Aloe Vera leaves under running water, followed by the removal of their outer skin. Subsequently, each leaf was divided into smaller pieces, from which the gel was allowed to seep out and carefully collected in a sterile container. The collected gel was then stored at 4°C until the time of its application in the study (adjunctive to SRP)
  Arms: scaling and root planing + 2.5% flurbiprofen on one site and 98% aloe vera on contralateral site; scaling and root planing + 98% aloe vera on one site and placebo on contralateral site
Other: Placebo — saline
  Arms: scaling and root planing + 2.5% flurbiprofen on one site and placebo on contralateral site; scaling and root planing + 98% aloe vera on one site and placebo on contralateral site

SUMMARY:
This study aims to evaluate clinically the efficacy of flurbiprofen gel in comparison to Aloe Vera gel as adjunctive to SRP in the reduction of periodontal pockets in patients with chronic periodontitis in smoking patients.

All patients will receive SRP prior to treatment.

* Group 1: one site will receive flurbiprofen while the contralateral site will receive a placebo
* Group 2: one site will receive aloe vera while the contralateral site will receive a placebo
* Group 3: one site will receive flurbiprofen while the contralateral site will receive aloe vera Researchers will compare the inter and intra-groups differences to check if there's a variation in the periodontal parameters measured.

DETAILED DESCRIPTION:
Complete medical and dental histories as well as informed consent will be collected from eligible participants, and periodontal charting will be done for them.

Medical history and laboratory screening for all patients will be carried out at baseline. All participants will undergo scaling and root planning. The selected patients will be allocated into three groups with the help of a computerized randomizer (Randomizer.org) and sites will be assigned as control or test based on a coin flip method:

* Group 1 (G1): 20 patients who received treatment involving the application of flurbiprofen gel as an adjunct to scaling and root planing. Specifically, on the test site of each patient, one milliliter of 2.5% flurbiprofen gel was applied, while on the contralateral side, placebo gel was administered as the control intervention.
* Group 2 (G2): 20 patients who received treatment involving the application of aloe Vera gel as an adjunct to scaling and root planing. Specifically, on the test site of each patient, one milliliter of 98% aloe Vera was applied, while on the contralateral side, placebo gel was administered as the control intervention.
* Group 3 (G3): The intervention involved applying flurbiprofen gel on one site, while the contralateral side received an application of 98% aloe vera.

The clinical examiner will not be informed of the treatment groups' distribution.

Patients will be informed on self-performed plaque control measures. In the 4th week, 8th week, 12th week, 6 months week clinical examination will be performed to measure the periodontal pocket depth, gingival index, plaque index, clinical attachment level (CAL),and bleeding on probing.

Statistical analysis was done using SAS 9.4 Software (SAS Institute Inc., Cary, NC, USA). Means and standard deviations (SD) were calculated for all continuous variables (periodontal parameters: CAL, PD, BOP, GI, PI) at the baseline, fourth week, eighth week, and twelfth week and 6 months. Repeated linear mixed-effects models (PROC MIXED in SAS) were used to examine the changes in all periodontal parameters over the five-time points within each group and between groups. An unstructured covariance matrix was used, residual plots were visually reviewed to check model fit, and extreme outliers were eliminated using the restricted likelihood distance. A Tukey-Kramer 8 correction was applied to all pairwise comparisons. One-way ANOVA was used to examine group differences in PD reduction and CAL. A p-value of 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion criteria: 60 patients were selected who had clinical periodontal loss and radiographic bone loss of stage III/grade C with no history of systemic disease. They had at least 2 periodontal sites with a pocket depth of six mm or greater, radiographic evidence of bone loss extending to the middle third of the root, and clinical attachment loss of five mm or more. Eligible subjects were categorized as current smokers if they consistently smoked more than 10 cigarettes per day for a minimum of 5 years. Additionally, individuals with no record of undergoing any periodontal treatment within the six months preceding the study were considered for inclusion.

Exclusion criteria: Patients with systemic illnesses such as diabetes mellitus or conditions that could potentially impair wound healing were excluded from participation. Additionally, individuals who were pregnant or lactating were not considered for inclusion in the study. Subjects who had been prescribed systemic antibiotics or non-steroidal anti-inflammatory drugs (NSAIDs) within the three months preceding the study were also excluded. Furthermore, individuals with confirmed or suspected hypersensitivity to Flurbiprofen or aloe Vera, the focus of the investigation, were not included in the study population.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-09-30 (Actual); Primary Completion 2023-05-25 (Actual); Study Completion 2023-07-19 (Actual)

PRIMARY OUTCOMES:
clinical attachment level | 6 months
  used to assess the loss of periodontal tissue support in periodontitis. It is the distance from the cemento-enamel junction (fixed point on the tooth) to the depth of the pocket
Probing Depth | 6 months
  used to detect the depth of the periodontal pocket. It is the distance from the gingival margin to the base of the pocket.

SECONDARY OUTCOMES:
Bleeding on Probing | 6 months
  It is an indicator of periodontal tissue inflammatory response. The probe is carefully introduced to the bottom of the pocket and gently moved laterally along the pocket wall. Depending on the severity of inflammation, bleeding can vary from a tenuous red line along the gingival sulcus to profuse bleeding (immediately after probing or few seconds after).
Plaque index | 6 months
  used to evaluate the level and rate of plaque formation on tooth surfaces. It measures the amount of dental plaque visible on the vestibular and lingual surfaces of all teeth, except the third molars. The amount of plaque is determined with disclosing solution and a range of scores of 0-5 is assigned with 0 denoting no plaque and 5 denoting heavy plaque (covering 2/3 of the tooth crown)
Gingival index | 6 months
  used to assess the severity of gingival inflammation. Scores ranges from 0-3 with 0 being normal and 3 being severe inflammation characterized by edema, redness, swelling, and spontaneous bleeding. This measurement is based on the presence or absence of bleeding on gentle probing

CONTACTS AND LOCATIONS:
Overall Officials: Nayer Aboelsaad, PhD, Study Chair — Professor and Chairman of Periodontology department - BeirutArabU
Locations (1):
- Beirut Arab University, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang S, Yu N, Arce RM. Periodontal inflammation: Integrating genes and dysbiosis. Periodontol 2000. 2020 Feb;82(1):129-142. doi: 10.1111/prd.12267. PMID 31850627
- [Background] Sanchavanakit N, Saengtong W, Manokawinchoke J, Pavasant P. TNF-alpha stimulates MMP-3 production via PGE2 signalling through the NF-kB and p38 MAPK pathway in a murine cementoblast cell line. Arch Oral Biol. 2015 Jul;60(7):1066-74. doi: 10.1016/j.archoralbio.2015.04.001. Epub 2015 Apr 20. PMID 25956994
- [Background] Offenbacher S, Farr DH, Goodson JM. Measurement of prostaglandin E in crevicular fluid. J Clin Periodontol. 1981 Aug;8(4):359-67. doi: 10.1111/j.1600-051x.1981.tb02045.x. PMID 7033302
- [Background] Khan KM, Kothari P, Du B, Dannenberg AJ, Falcone DJ. Matrix metalloproteinase-dependent microsomal prostaglandin E synthase-1 expression in macrophages: role of TNF-alpha and the EP4 prostanoid receptor. J Immunol. 2012 Feb 15;188(4):1970-80. doi: 10.4049/jimmunol.1102383. Epub 2012 Jan 6. PMID 22227567
- [Background] Eke PI, Wei L, Thornton-Evans GO, Borrell LN, Borgnakke WS, Dye B, Genco RJ. Risk Indicators for Periodontitis in US Adults: NHANES 2009 to 2012. J Periodontol. 2016 Oct;87(10):1174-85. doi: 10.1902/jop.2016.160013. Epub 2016 Jul 1. PMID 27367420
- [Background] Kim J, Amar S. Periodontal disease and systemic conditions: a bidirectional relationship. Odontology. 2006 Sep;94(1):10-21. doi: 10.1007/s10266-006-0060-6. PMID 16998613
- [Background] Ehizele A, Akhionbare O. Effect of non-surgical periodontal therapy on the concentration of volatile sulfur compound in mouth air of a group of nigerian young adults. Ann Med Health Sci Res. 2013 Jul;3(3):433-7. doi: 10.4103/2141-9248.117951. PMID 24116328
- [Background] Choi YM, Lee JY, Choi J, Joo JY. Effect of root planing on the reduction of probing depth and the gain of clinical attachment depending on the mode of interproximal bone resorption. J Periodontal Implant Sci. 2015 Oct;45(5):184-9. doi: 10.5051/jpis.2015.45.5.184. Epub 2015 Nov 2. PMID 26550527
- [Background] Morozumi T, Kubota T, Abe D, Shimizu T, Nohno K, Yoshie H. Microbiological effect of essential oils in combination with subgingival ultrasonic instrumentation and mouth rinsing in chronic periodontitis patients. Int J Dent. 2013;2013:146479. doi: 10.1155/2013/146479. Epub 2013 Sep 19. PMID 24171000
- [Background] Goodson JM, Dewhirst FE, Brunetti A. Prostaglandin E2 levels and human periodontal disease. Prostaglandins. 1974 Apr 10;6(1):81-5. doi: 10.1016/s0090-6980(74)80043-2. No abstract available. PMID 4595580
- [Background] Bacchi S, Palumbo P, Sponta A, Coppolino MF. Clinical pharmacology of non-steroidal anti-inflammatory drugs: a review. Antiinflamm Antiallergy Agents Med Chem. 2012;11(1):52-64. doi: 10.2174/187152312803476255. PMID 22934743
- [Background] Ren J, Fok MR, Zhang Y, Han B, Lin Y. The role of non-steroidal anti-inflammatory drugs as adjuncts to periodontal treatment and in periodontal regeneration. J Transl Med. 2023 Feb 25;21(1):149. doi: 10.1186/s12967-023-03990-2. PMID 36829232
- [Background] Marcum ZA, Hanlon JT. Recognizing the Risks of Chronic Nonsteroidal Anti-Inflammatory Drug Use in Older Adults. Ann Longterm Care. 2010;18(9):24-27. PMID 21857795
- [Background] Sholapurkar A, Sharma D, Glass B, Miller C, Nimmo A, Jennings E. Professionally Delivered Local Antimicrobials in the Treatment of Patients with Periodontitis-A Narrative Review. Dent J (Basel). 2020 Dec 22;9(1):2. doi: 10.3390/dj9010002. PMID 33375176
- [Background] Salvi GE, Lang NP. The effects of non-steroidal anti-inflammatory drugs (selective and non-selective) on the treatment of periodontal diseases. Curr Pharm Des. 2005;11(14):1757-69. doi: 10.2174/1381612053764878. PMID 15892673
- [Background] Howell TH, Fiorellini J, Weber HP, Williams RC. Effect of the NSAID piroxicam, topically administered, on the development of gingivitis in beagle dogs. J Periodontal Res. 1991 May;26(3 Pt 1):180-3. doi: 10.1111/j.1600-0765.1991.tb01643.x. PMID 1830620
- [Background] Deshpande NC, Bhat KM, Bhat GS, Deshpande AN. Randomized, controlled clinical study to evaluate efficacy of novel indigenously designed controlled release flurbiprofen gel system for management of periodontal diseases. Contemp Clin Dent. 2013 Jan;4(1):32-6. doi: 10.4103/0976-237X.111591. PMID 23853449
- [Background] Saglam M, Kantarci A, Dundar N, Hakki SS. Clinical and biochemical effects of diode laser as an adjunct to nonsurgical treatment of chronic periodontitis: a randomized, controlled clinical trial. Lasers Med Sci. 2014 Jan;29(1):37-46. doi: 10.1007/s10103-012-1230-0. Epub 2012 Nov 16. PMID 23161345
- [Background] Pradeep AR, Bajaj P, Agarwal E, Rao NS, Naik SB, Kalra N, Priyanka N. Local drug delivery of 0.5% azithromycin in the treatment of chronic periodontitis among smokers. Aust Dent J. 2013 Mar;58(1):34-40. doi: 10.1111/adj.12019. Epub 2013 Jan 30. PMID 23441790
- [Background] Agarwal E, Pradeep AR, Bajaj P, Naik SB. Efficacy of local drug delivery of 0.5% clarithromycin gel as an adjunct to non-surgical periodontal therapy in the treatment of current smokers with chronic periodontitis: a randomized controlled clinical trial. J Periodontol. 2012 Sep;83(9):1155-63. doi: 10.1902/jop.2012.110600. Epub 2012 Jan 16. PMID 22248223
- [Background] Eick S, Renatus A, Heinicke M, Pfister W, Stratul SI, Jentsch H. Hyaluronic Acid as an adjunct after scaling and root planing: a prospective randomized clinical trial. J Periodontol. 2013 Jul;84(7):941-9. doi: 10.1902/jop.2012.120269. Epub 2012 Oct 22. PMID 23088524
- [Background] Prasad D, Kunnaiah R. Punica granatum: A review on its potential role in treating periodontal disease. J Indian Soc Periodontol. 2014 Jul;18(4):428-32. doi: 10.4103/0972-124X.138678. PMID 25210254
- [Background] Krayer JW, Leite RS, Kirkwood KL. Non-surgical chemotherapeutic treatment strategies for the management of periodontal diseases. Dent Clin North Am. 2010 Jan;54(1):13-33. doi: 10.1016/j.cden.2009.08.010. PMID 20103470
- [Background] Eid Abdelmagyd HA, Ram Shetty DS, Musa Musleh Al-Ahmari DM. Herbal medicine as adjunct in periodontal therapies- A review of clinical trials in past decade. J Oral Biol Craniofac Res. 2019 Jul-Sep;9(3):212-217. doi: 10.1016/j.jobcr.2019.05.001. Epub 2019 May 14. PMID 31193290
- [Background] Taleghani F, Rezvani G, Birjandi M, Valizadeh M. Impact of green tea intake on clinical improvement in chronic periodontitis: A randomized clinical trial. J Stomatol Oral Maxillofac Surg. 2018 Nov;119(5):365-368. doi: 10.1016/j.jormas.2018.04.010. Epub 2018 Apr 30. PMID 29723659
- [Background] Mekhemar M, Geib M, Kumar M, Radha, Hassan Y, Dorfer C. Salvadora persica: Nature's Gift for Periodontal Health. Antioxidants (Basel). 2021 Apr 30;10(5):712. doi: 10.3390/antiox10050712. PMID 33946353
- [Background] Vogler BK, Ernst E. Aloe vera: a systematic review of its clinical effectiveness. Br J Gen Pract. 1999 Oct;49(447):823-8. PMID 10885091
- [Background] Harlev E, Nevo E, Lansky EP, Ofir R, Bishayee A. Anticancer potential of aloes: antioxidant, antiproliferative, and immunostimulatory attributes. Planta Med. 2012 Jun;78(9):843-52. doi: 10.1055/s-0031-1298453. Epub 2012 Apr 19. PMID 22516934
- [Background] Pareek S, Nagaraj A, Sharma P, Atri M, Walia S, Naidu S, Yousuf A. Disinfection of dental unit water line using aloe vera: in vitro study. Int J Dent. 2013;2013:618962. doi: 10.1155/2013/618962. Epub 2013 Sep 8. PMID 24089615
- [Background] Im SA, Kim KH, Kim HS, Lee KH, Shin E, Do SG, Jo TH, Park YI, Lee CK. Processed Aloe vera gel ameliorates cyclophosphamide-induced immunotoxicity. Int J Mol Sci. 2014 Oct 24;15(11):19342-54. doi: 10.3390/ijms151119342. PMID 25347273
- [Background] Athiban PP, Borthakur BJ, Ganesan S, Swathika B. Evaluation of antimicrobial efficacy of Aloe vera and its effectiveness in decontaminating gutta percha cones. J Conserv Dent. 2012 Jul;15(3):246-8. doi: 10.4103/0972-0707.97949. PMID 22876011
- [Background] Doddanna SJ, Patel S, Sundarrao MA, Veerabhadrappa RS. Antimicrobial activity of plant extracts on Candida albicans: an in vitro study. Indian J Dent Res. 2013 Jul-Aug;24(4):401-5. doi: 10.4103/0970-9290.118358. PMID 24047829
- [Background] Babaee N, Zabihi E, Mohseni S, Moghadamnia AA. Evaluation of the therapeutic effects of Aloe vera gel on minor recurrent aphthous stomatitis. Dent Res J (Isfahan). 2012 Jul;9(4):381-5. PMID 23162576
- [Background] Pradeep AR, Agarwal E, Naik SB. Clinical and microbiologic effects of commercially available dentifrice containing aloe vera: a randomized controlled clinical trial. J Periodontol. 2012 Jun;83(6):797-804. doi: 10.1902/jop.2011.110371. Epub 2011 Nov 16. PMID 22087805
- [Background] Namiranian H, Serino G. The effect of a toothpaste containing aloe vera on established gingivitis. Swed Dent J. 2012;36(4):179-85. PMID 23421308
- [Background] Chandrahas B, Jayakumar A, Naveen A, Butchibabu K, Reddy PK, Muralikrishna T. A randomized, double-blind clinical study to assess the antiplaque and antigingivitis efficacy of Aloe vera mouth rinse. J Indian Soc Periodontol. 2012 Oct;16(4):543-8. doi: 10.4103/0972-124X.106905. PMID 23493442
- [Background] Ashouri Moghaddam A, Radafshar G, Jahandideh Y, Kakaei N. Clinical Evaluation of Effects of Local Application of Aloe vera Gel as an Adjunct to Scaling and Root Planning in Patients with Chronic Periodontitis. J Dent (Shiraz). 2017 Sep;18(3):165-172. PMID 29034270
- [Background] Nayer Aboelsaad, et al. (2014) Clinical Efficacy of Local Delivered Minocycline in the Treatment of Chronic Periodontitis Smoker Patients. J Dent Oral Health 1: 1-5
- [Background] Brad W. Neville DDS, ... Angela C. Chi DMD, in Color Atlas of Oral and Maxillofacial Diseases, 2019

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-09-30): https://cdn.clinicaltrials.gov/large-docs/78/NCT06041178/Prot_SAP_000.pdf
  • Informed Consent Form (2022-09-30): https://cdn.clinicaltrials.gov/large-docs/78/NCT06041178/ICF_001.pdf